CLINICAL TRIAL: NCT05692791
Title: The Relationship Between Two-point Discrimination and Position Perception in Children Who Have Idiopathic Toe Walk
Brief Title: Idiopathic Toe-Walking Position Sensation
Status: Completed | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Ömer Faruk ÖZÇELEP, Lecturer, Kirsehir Ahi Evran Universitesi
Other Study IDs: AEUnivers
Record Dates: First submitted 2023-01-12; First posted 2023-01-20 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Gait Disorder, Sensorimotor
Keywords: Idiopathic Toe Walking
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ITW
  Interventions: Diagnostic Test: Two-point Discrimination Test; Diagnostic Test: Semmes-Weinstein monofilament test
- Control Group
  Interventions: Diagnostic Test: Two-point Discrimination Test; Diagnostic Test: Semmes-Weinstein monofilament test

INTERVENTIONS:
Diagnostic Test: Two-point Discrimination Test — Two-point discrimination (2PD) is the ability to discern that two nearby objects touching the skin are truly two distinct points, not one. It is often tested with two sharp points during a neurological examination and is assumed to reflect how finely innervated an area of skin is.
Diagnostic Test: Semmes-Weinstein monofilament test — Semmes-Weinstein monofilament test is used to assess light touch sensations.

SUMMARY:
The aim of this study is to investigate the effect of plantar two-point discrimination on hip-knee-ankle position sense in children with toe walking.The main questions it aims to answer are:

* Are two-point discrimination and light pressure sensation in the plantar region affected in children with idiopathic toe gait?
* Does the two-point discrimination in the plantar in general and the heel in particular affect the position sense of the hip-knee and ankle?

DETAILED DESCRIPTION:
Children who tend to walk on toes after they should have developed a heel-toe gait are diagnosed with idiopathic toe walking (ITW).Cerebral palsy, muscular dystrophy, and orthopaedic problems such congenital talipes equinus are some of the diseases that are frequently linked to a toe-walking gait. A diagnosis of ITW is made when there is no physical or medical cause for the absence of a heel strike. Five percent of healthy children are estimated to have ITW, and boys are more likely than girls to be affected. Reduced ankle range of motion is prevalent symptom in children with ITW. Since ITW often manifests as symmetrical tiptoe walking in children, reports showing a comparable bilateral reduction in ankle range of motion at both lower limbs indicate the symmetrical character of this gait type. Lower vibration perception thresholds, a tendency to be left-handed, and noticeable variations in sensory seeking and modulation scores are all characteristics of children with an ITW gait.

The small fibers that innervate the cutaneous receptors (such as Merkel's cell, Pacinian corpuscles, Meissner's corpuscles, and Ruffini endings in the skin) are more crucial for postural control than the large fibers that innervate the major muscle spindles and the Golgi tendon organs. Standing balance control is more dependent on Merkel's cells and Ruffini endings (slow adapting receptors), which are in charge of touch and pressure sensitivity, than it is on Meissner's and Pacinian corpuscles (rapid adapting receptors), which are in charge of vibrotactile sensitivity.Additionally, it has been demonstrated that tactile sensation in the foot sole affects the activity of the tibialis anterior muscle as well as the regulation of gait pattern at lower limb joints. These investigations support the notion that cutaneous feeling is crucial for preserving postural and gait stability.The literature states that plantar pressure and sensory changes have disruptive effects on postural control.The aim of this study is to investigate the effect of plantar two-point discrimination on hip-knee-ankle position sense in children with toe walking.

ELIGIBILITY:
Inclusion Criteria:

* Having idiopathic toe walking diagnosis

Exclusion Criteria:

* Having another known neuromuscular disease

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children who have idiopathic toe walking in the experimental group and healthy children in the control group with the same ages.
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Hip-Knee-Ankle Joint Position Sense | 15 weeks
  Position the body segment being tested and then passively position the individual's joint in space. Hold the lateral surfaces of the limb to minimize cues from touch and pressure sensations.
  Move the body segment into a position and either have the patient maintain the position or assist the patient in maintaining the position if needed.
  Have the patient duplicate the position with the opposite extremity. The procedure is repeated enough times to conclude if joint position sense is intact or impaired. A suggested minimum number of trials is five per joint.

CONTACTS AND LOCATIONS:
Locations (1):
- Ahi Evran University, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
With mail
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months after publishing

REFERENCES:
- [Background] Silva PG, Jones A, Araujo PM, Natour J. Assessment of light touch sensation in the hands of systemic sclerosis patients. Clinics (Sao Paulo). 2014 Sep;69(9):585-8. doi: 10.6061/clinics/2014(09)02. PMID 25318088
- [Background] Westberry DE, Davids JR, Davis RB, de Morais Filho MC. Idiopathic toe walking: a kinematic and kinetic profile. J Pediatr Orthop. 2008 Apr-May;28(3):352-8. doi: 10.1097/BPO.0b013e318168d996. PMID 18362803